CLINICAL TRIAL: NCT02882633
Title: Lumbar Plexus Block vs Fascia Iliaca Block After Hip Arthroscopy: A Non-inferiority Study
Brief Title: Lumbar Plexus Block vs Fascia Iliaca Block After Hip Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 822547Upenn
Record Dates: First submitted 2016-08-16; First posted 2016-08-30 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Hip Arthroscopy; Nerve Block
Keywords: lumbar plexus block; fascia iliac block; quality of recovery score; pain score
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumbar Plexus Block (Active Comparator): Subjects will receive single shot local anesthetic, 30 ml bolus of bupivacaine, given preoperatively to help with postoperative pain
  Interventions: Drug: 30ml bolus of bupivacaine
- Fascia Iliac Block (Active Comparator): Subjects will receive single shot local anesthetic, 30 ml bolus of bupivacaine, given preoperatively to help with postoperative pain
  Interventions: Drug: 30ml bolus of bupivacaine

INTERVENTIONS:
Drug: 30ml bolus of bupivacaine — Local anesthetic
  Other Names: Marcaine; Sensorcaine

SUMMARY:
The purpose of this study is to compare lumbar plexus block to fascia iliac block done in adult patients who have undergone hip arthroscopy surgery. Visual analogue scores, opioid consumption, and quality of recovery 48 hours post operatively will be used for comparison.

DETAILED DESCRIPTION:
If the patient is willing to participate and signs the consent, he/she will be randomized to one of the two treatment groups:

1. Lumbar Plexus Block
2. Fascia Iliaca Block

The patient will undergo general anesthesia as by the attending anesthesiologist assigned to the case. No intraoperative restrictions will be required for this study. Once in the PACU, the patient will be assessed and if their pain score is ≥ 4 on the NRS, the patient will be randomized to a lumbar plexus block or fascia iliaca block.

Patients will be monitored during block performance with standard ASA monitors. All patients will receive 2 L of oxygen via a nasal cannula. Sedatives will be titrated to effect. Midazolam 1-2 mg, and fentanyl 50-100 mcg will be used for sedation.

The fascia iliaca block will be performed in a standard fashion as described2. The patient will be placed in a supine position. The ipsilateral groin will be prepped and cleaned with chlorhexidine. An ultrasound machine with a linear transducer covered with a sterile tegaderm will be utilized. The transducer is placed inferior to the inguinal ligament until the femoral artery is located. The probe is then moved laterally until the Sartorius muscle is seen. A skin wheal with 3ml of 1% lidocaine is made and a 2-inch blunt tip needle is inserted in plane. The needle is seen to pierce the fascia iliaca and 1-2 ml of 0.25% Preservative Free bupivacaine with 1:200,000 epinephrine is injected to confirm correct needle placement between the fascia iliaca and iliopsoas muscle. An injection will be deemed adequate if local anesthetic is seen to separate these two layers in a medial to lateral direction. A total of 30ml of the above solution will be injected.

The lumbar plexus block will be performed with the patient placed in a lateral position with the operative side facing up. An ultrasound machine with a curved transducer covered with a sterile tegaderm will be utilized. The ipsilateral hip and knee will be flexed to 90 degrees. The anatomy for the LP block will be localized using a modified transverse scan of the lumbar paravertebral area (PMTS). This technique is well described by Karmarkar et al.7 The target vertebral level will be identified by locating the lumbosacral junction (the gap of L5-S1) using a paramedian sagittal scan and then counting cranially to locate both the lamina and the transverse process of L3-L5. The transducer is then placed 4 cm lateral to the midline at the L3-4 level and directed medially to insonate the intervertebral foramen through the lumbar intervertebral space. A skin wheal is made at this site with 1% lidocaine. and a 4 inch blunt tip needle is introduced 4 cm lateral to the midline and just medial of the transducer after connecting it to a nerve stimulator set at 1.00 mA. The needle is slowly advanced under ultrasound guidance until engaged in the psoas compartment and a quadriceps twitch is elicited. The nerve stimulator is turned down until the twitch is abolished at 0.3mA or less. 1-2cmlof 0.25% Preservative free Bupivacaine with 1:200,000 epinephrine is injected slowly after negative aspiration. A total of 30ml will be injected. Spread will be confirmed with ultrasound.

All patients will receive prophylaxis for postoperative nausea and vomiting (PONV) during surgery. The protocol for prophylaxis against PONV includes administration of 4 mg of dexamethasone after induction of anesthesia and 4 mg of ondansetron 20 minutes before recovery from anesthesia. Dexamethasone is withheld if the patient has poorly controlled diabetes mellitus (DM). Uncontrolled DM will be defined as random blood glucose above 250 mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients18 years and older scheduled for hip arthroscopy surgery
* American Society of Anesthesiologists (ASA) physical status I -III
* Mentally competent and able to give consent for enrollment in the study

Exclusion Criteria:

* Chronic opioid use (use of any opioid daily or on most days of the week for more than 3 months)
* Diagnosed peripheral neuropathy in the surgical lower extremity
* Allergy to study medications
* BMI >42

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-11; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Badiola, MD, Principal Investigator — Univeristy of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lumbar Plexus Block | Fascia Iliac Block
Started | 25 | 25
Completed | 23 | 25
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fascia Iliaca Block: Subjects will receive single shot local anesthetic, 30 ml bolus of bupivacaine, given preoperatively to help with postoperative pain
  30ml bolus of bupivacaine: Local anesthetic
- Total: Total of all reporting groups
Arm/Group | Lumbar Plexus Block | Fascia Iliaca Block | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.83 (11.55) | 39.8 (11.40) | 39.34 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 7 | 9 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.89 (6.59) | 26.80 (4.52) | 28.28 (5.76)
Femoral/Acetabular osteoplasty [Count of Participants; unit: Participants] | 19 | 23 | 42
Peri-trochanteric space surgery [Count of Participants; unit: Participants] | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Change
Description: Change in pain scores, as measured by the Visual Analog Scale (0-10). 10 is worst imaginable pain and 0 means no pain at all.
Time Frame: Change from baseline through 15 minutes
Measure: Mean (Inter-Quartile Range); unit: change in score on a scale
Arm/Group | Lumbar Plexus Block | Fascia Iliac Block
Number analyzed (Participants) | 23 | 25
change in score on a scale | 3 [1 to 3] | 1.72 [0 to 8]

2. Primary Outcome: Amount of Opiate Consumption
Description: Participants need for pain relief as measured by opiate consumption
Time Frame: While in PACU. An average length of stay for Lumbar Plexus Block group was 165.04 min and 139.72 min for Fascia Iliaca Block group.
Measure: Mean (Inter-Quartile Range); unit: mg
Arm/Group | Lumbar Plexus Block | Fascia Iliac Block
Number analyzed (Participants) | 23 | 25
mg | 16.98 [5.81 to 22.5] | 20.80 [5.62 to 33.75]

3. Secondary Outcome: Quality of Recovery
Description: Score of QoR survey to determine recovery status. 0-18 where 0 is the worst and 18 is the best feeling.
Time Frame: Change from baseline through 24 hours
Measure: Mean (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Lumbar Plexus Block | Fascia Iliac Block
Number analyzed (Participants) | 23 | 25
Score on a scale | 14.52 [14 to 17] | 15.91 [11 to 18]

ADVERSE EVENTS:
Time Frame: Adverse Effects data collected day of procedure and following 48 hours
Arm/Group | Lumbar Plexus Block | Fascia Iliac Block
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/25
Other Adverse Events (participants affected / at risk) | 1/23 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumbar Plexus Block (N=23) | Fascia Iliac Block (N=25)
Epidural Spread (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumbar Plexus Block (N=23) | Fascia Iliac Block (N=25)
Epidural Spread (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT02882633/Prot_SAP_000.pdf